CLINICAL TRIAL: NCT02728180
Title: Xingnaojing for Moderate-to-severe Acute Ischemic Stroke (XMAS): A Multicenter, Prospective, Randomized, Open-label, Blinded Endpoint Clinical Trial.
Brief Title: Xingnaojing for Moderate-to-severe Acute Ischemic Stroke (XMAS)
Acronym: XMAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Chao Yang Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Beijing Emergency Medical Center (Other); Chengdu University of Traditional Chinese Medicine (Other); Deyang People's Hospital (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Hunan Academy of Chinese Medicine (Unknown); The First Hospital of Jilin University (Other); China-Japan Union Hospital, Jilin University (Other); Jiangmen Wuyi Hospital of Traditional Chinese Medicine (Other); Jiangxi Provincial People's Hopital (Other); Mianyang Central Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shandong University of Traditional Chinese Medicine (Other); Shaanxi Provincial People's Hospital (Other); Shaanxi Provincial Hospital of Traditional Chinese Medicine (Unknown); The Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown); Tianshui Hospital of Traditional Chinese Medicine (Unknown); Wuxi Hospital of Traditional Chinese Medicine (Unknown); The First Hospital of Wuhan (Unknown); Zhejiang Provincial Tongde Hospital (Other); Zhejiang Provincial Hospital of TCM (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); The Fifth People Hospital of Chongqing (Unknown); Chongqing Traditional Chinese Medicine Hospital (Other); Zibo Hospital of Traditional Chinese Medicine (Other); Liling Hospital of Traditional Chinese Medicine (Unknown); Cangzhou Hospital of Integrated Medicine (Unknown); Yantai Yuhuangding Hospital (Other)
Responsible Party: Principal Investigator, Ying Gao, Vice president of Dongzhimen Hospital, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014BAI10B05-01
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Xingnaojing injection; Randomized Controlled Trial; Traditional Chinese Medicine
MeSH Terms: conditions — Ischemic Stroke | interventions — xingnaojing; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xingnaojing and standard care (Experimental): Subjects will receive intravenously administered Xingnaojing injection, combined with guidelines-based standard care.
  Interventions: Drug: Xingnaojing injection; Other: Standard care
- Standard care only (Active Comparator): Subjects will receive guidelines-based standard care only.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Xingnaojing injection — Xingnaojing injection (20 ml), IV (in the vein), every 12 hours for 10 days.
  Arms: Xingnaojing and standard care
Other: Standard care — Guidelines-based standard care for acute ischemic stroke.

SUMMARY:
The main purpose of this trial is to determine whether Xingnaojing, intravenously administered within 24 hours of symptom onset, improves the 3-month outcome in participants with acute ischemic stroke.

DETAILED DESCRIPTION:
Xingnaojing is widely used in China, but there is lack of high-quality evidence of its efficacy for acute ischemic stroke currently. The primary hypothesis of this trial is that Xingnaojing will increase the proportion of people alive and independent at three months. Xingnaojing, combined with guidelines-based standard care, will be compared to standard care alone in patients with acute ischemic stroke within 24 hours of symptom onset. All patients will have a National Institutes of Health Stroke Scale (NIHSS) entry score of 5-20. Patients in each group will be treated according to the guidelines-based standard care, including intravenous thrombolysis if appropriate. The primary outcome will be determined at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within 24 hours of symptom onset.
* National Institutes of Health Stroke Scale score ≥ 5 and ≤ 20.
* Age ≥ 35 and ≤ 80 years.
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Planned or already received endovascular treatment.
* Suspected secondary stroke caused by tumor, brain trauma, or hematologic diseases.
* Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scare score ≥2 ).
* Other conditions that lead to motor dysfunction (e.g. severe osteoarthrosis, rheumatoid arthritis).
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase, or aspartate aminotransferase value that is twice greater than the upper limit of normal).
* Life expectancy of 90 days or less due to other life threatening illness (e.g. advanced cancer).
* Other conditions that render outcomes or follow-up unlikely to be assessed..
* Known to be pregnant or breastfeeding.
* Currently receiving an investigational drug.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients independent | 90 days
  Proportion of patients independent is defined as Modified Rankin Scale score of 0, 1, or 2.

SECONDARY OUTCOMES:
Comparison of the change in the NIHSS scores from baseline to 10 days in the two groups. | Baseline and 10 days.
  The NIHSS score ranges from 0 (best score) to 42 (worst score).
Activities of daily living | 30 days and 90 days
  Activities of daily living measured by Barthel Index score at 30 days and 90 days.
Patient reported outcome (PRO) scale of stroke | 10 days
  Patient reported outcome (PRO) scale of stroke at 10 days.
Early neurologic deterioration (END) | Baseline and 48 hours
  Early neurologic deterioration is defined as an increase of 3 points or more in the NIHSS score between baseline and 48 hours.
Symptomatic Intracranial Hemorrhage (sICH) | 10 dyas
  Symptomatic Intracranial Hemorrhage (sICH) within 10 days of stroke onset. (Any ICH related to a decline in neurologic status or the development of new neurologic symptoms which in the judgment of the clinical investigator was related to the ICH.)
Deaths from any cause | 10 days, 90 days
  Number of deaths from any cause within 10 days and 90 days after symptom onset.
Safety end points - Number of patients with any adverse events, results of electrocardiography, vital signs and laboratory tests (complete blood count, chemistry and urinalysis). | 10 days
  Number of patients with any adverse events, results of electrocardiography, vital signs and laboratory tests (complete blood count, chemistry and urinalysis).
Cardiovascular events | 90 days
  Number of patients with recurrence of stroke or myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lai X, Cao K, Kong L, Liu Q, Gao Y; XMAS study investigators. Xingnaojing for Moderate-to-severe Acute ischemic Stroke (XMAS): study protocol for a randomized controlled trial. Trials. 2017 Oct 16;18(1):479. doi: 10.1186/s13063-017-2222-y. PMID 29037226